CLINICAL TRIAL: NCT05213182
Title: Community-Based Peer Support Intervention to Mitigate Social Isolation and Stigma of Adolescent Motherhood in Harare, Zimbabwe
Brief Title: Peer Support Intervention to Mitigate Social Isolation and Stigma of Adolescent Motherhood in Zimbabwe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West Chester University of Pennsylvania (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of South Carolina (Other); Organization for Public Health Interventions and Development (Unknown); University of Zimbabwe (Other); SpeakUp! Pennsylvania (Unknown)
Responsible Party: Principal Investigator, Chiwoneso Tinago, Associate Professor, West Chester University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20180723A
Record Dates: First submitted 2022-01-05; First posted 2022-01-28 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Mental Health Disorder; Social Isolation; Stigma, Social
Keywords: Adolescent Mothers; Mental Health; Social Isolation; Stigma; Zimbabwe; Peer Support; WhatsApp Messenger
MeSH Terms: conditions — Mental Disorders; Social Isolation; Social Stigma; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A quasi-experimental design was used, and the research tested differential changes over base-, mid-, and end-line in mental health and social support outcomes among adolescent mothers (14-18 years) in the intervention and control arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm (n=104 adolescent mothers) participated in the 12 in-person peer support group sessions and completed sociodemographic, base-, mid-, and end-line surveys.
  Interventions: Behavioral: Young Women of Today
- Control (No Intervention): The control arm (n=79 adolescent mothers) completed sociodemographic, base-, mid- and end-line surveys.

INTERVENTIONS:
Behavioral: Young Women of Today — Adolescent mothers engaged in the development and implementation of the intervention which also involved key community stakeholders to address stigma related to mental illness and adolescent motherhood. Community health workers and peer educators in the intervention arm were recruited and trained on co-facilitating peer support groups. The intervention arm (n=104 adolescent mothers) participated in the peer support groups and completed sociodemographic, base-, mid-, and end-line surveys. The control arm (n=79 adolescent mothers) completed sociodemographic, base-, mid- and end-line surveys. Peer support groups (12 groups with 6-12 participants in each group) met in-person twice a month and completed 12 peer-group sessions from May-August 2019 addressing participant identified topics such as depression. WhatsApp Messenger was used for training and implementation support. Key community stakeholders met to discuss project progress and recommendations to improve adolescent mothers' health.
  Other Names: Community-based Peer Support Intervention to Mitigate Social Isolation and Stigma of Adolescent Motherhood in Harare, Zimbabwe
  Arms: Intervention

SUMMARY:
A community-based peer support intervention for adolescent mothers aged 14-18 years in Harare, Zimbabwe was developed and tested in partnership with adolescent mothers, community health workers, and key community stakeholders. The intervention leveraged peer support, technology via WhatsApp Messenger, community health workers, peer educators and involvement of key community stakeholders to reduce prevalence of loneliness, depressive symptoms and common mental disorders, improve perceived social support, and develop coping, parenting, and communication skills to mitigate potential stressors and stigma of adolescent motherhood.

DETAILED DESCRIPTION:
Adolescent mothers in Zimbabwe often experience stigma and feel isolated due to lack of social support with a loss of social networks and educational opportunities. Adolescent mothers may also lack coping skills and resources to successfully navigate motherhood. Unless addressed, these circumstances may have negative consequences for the mental health of the adolescent mother and downstream consequences for their children. A quasi-experimental design was used, and the research tested differential changes over base-, mid-, and end-line in mental health and social support outcomes among adolescent mothers (14-18 years) in the intervention and control arms. The study addressed two objectives:

1. Understand and describe perceptions and experiences with adolescent motherhood and their influence on health.
2. Explore the acceptability and effectiveness of a community-based peer support intervention for adolescent mothers in a high-density low-income community in Harare to mitigate potential stressors and stigma of adolescent motherhood.

Adolescent mothers engaged as active participants in the development (e.g., defining their needs) and implementation of the intervention which also involved key community stakeholders to address stigma related to mental illness and adolescent motherhood. Existing community resources were leveraged such as peer support, health workers, and technology through WhatsApp Messenger, a popular and low-cost messaging app, to deliver some intervention components and as a platform for communication and training support for peer support group facilitators. Community health workers and peer educators in the intervention arm were recruited and trained on co-facilitating peer support groups. The intervention arm (n=104 adolescent mothers) participated in the peer support groups and completed sociodemographic, base-, mid-, and end-line surveys. The control arm (n=79 adolescent mothers) completed sociodemographic, base-, mid- and end-line surveys. Peer support groups (12 groups with 6-12 participants in each group) met in-person twice a month and completed 12 peer-group sessions from May-August 2019 addressing participant identified topics such as income generation, depression, and healthy parenting. WhatsApp Messenger was used for training and implementation support. Key community stakeholders met to discuss project progress and recommendations to improve the health of adolescent mothers. Data were analyzed using Stata 13 software.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent mothers (pregnant and/or have a child or children) aged 14-18 years living in the intervention or control communities.

Exclusion Criteria:

* Individuals who are not adolescent mothers aged 14-18 years and who do not live in the intervention or control communities.
* individuals with an acute or severe illness or disability (e.g. psychosis) that results in a functional impairment that substantially interferes with the ability to provide informed consent and participate in the study.

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants who identified as adolescent mothers (pregnant and/or have a child or children) aged 14-18 years.
Enrollment: 183 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms and Suicidal Ideation | 6 months
  Change from baseline to endline in depressive symptoms and suicide ideation using the Patient Health Questionnaire, a validated 9-item tool utilized to screen, diagnose, monitor, and measure depression severity and suicide ideation. The scoring of the questionnaire is as follows: 0-4 minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, 20-27 severe depression. Thus higher scores mean a worse outcome.
Perceived Social Support | 6 months
  Change from baseline to endline in perceived social support using the Multidimensional Scale of Perceived Social Support a validated scale that measures perceived social support among participants' friends, family and significant others.This scale has 12 items used to assess social support using a Likert scale. The scale measures social support from three categories: family, friends, and significant other. Results ranging from 1 to 2.9 could be considered low support; a score of 3 to 5 could be considered moderate support; a score from 5.1 to 7 could be considered high support. Thus higher scores mean a better outcome.

SECONDARY OUTCOMES:
Common Mental Disorders | 6 months
  Change from baseline to endline in common mental disorders using the 14-item Shona Symptom Questionnaire, a culturally appropriate common mental disorders screening tool. Participants scoring 7 or below are defined as not having a common mental disorder. Participants scoring 8 or more are defined as having a common mental disorder. Thus higher scores mean a worse outcome.
Peer and Significant Adult Support | 6 months
  Change from baseline to endline in peer and significant adult support using the Peer and Significant Adult Support Survey, which was developed by the research team. Using a Likert scale of 0 (not at all), 1 (some of the time), 2 (most of the time), and 3 (all the time) to measure perceived social support from peers and significant adults, a higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Chiwoneso Tinago, PhD, Principal Investigator — West Chester University of Pennsylvania
Locations (1):
- West Chester University of Pennsylvania, West Chester, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tinago CB, Frongillo EA, Warren AM, Chitiyo V, Jackson TN, Cifarelli AK, Fyalkowski S, Pauline V. Testing the Effectiveness of a Community-Based Peer Support Intervention to Mitigate Social Isolation and Stigma of Adolescent Motherhood in Zimbabwe. Matern Child Health J. 2024 Apr;28(4):657-666. doi: 10.1007/s10995-023-03821-2. Epub 2023 Nov 13. PMID 37957412